CLINICAL TRIAL: NCT04015037
Title: Double-blind Randomized Study on the Effect of Non-hormonal Gel Application to the Genital Area of Women in the Menacme With Sexual Dysfunction
Brief Title: The Effect of Non-hormonal Gel Application in Women in the Menacme With Sexual Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JULIANA AQUINO DE MOURA (Other)
Responsible Party: Sponsor-Investigator, JULIANA AQUINO DE MOURA, Principal Investigator, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 933.092
Record Dates: First submitted 2017-11-29; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: Randomized double-blind placebo-controlled study with women with age greater than 20, in the menacme, with complaints about sexual activity.
Who Masked: Participant, Investigator
Masking Description: The party or parties involved in the clinical trial who are prevented from having knowledge of the interventions assigned to individual participants. Select all that apply.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The participants will be with age greater than 20 old, be in either the menacme (not pregnant). They will have complaints about sexual activity, an active sex life, and body mass index (BMI) equal to or less than 30. Through these criteria of inclusion and exclusion
  Interventions: Combination Product: placebo or drug
- Group B (Experimental): The participants will be with age greater than 20 old, be in either the menacme (not pregnant). They will have complaints about sexual activity, an active sex life, and body mass index (BMI) equal to or less than 30. Through these criteria of inclusion and exclusion
  Interventions: Combination Product: placebo or drug

INTERVENTIONS:
Combination Product: placebo or drug — Group A and B (medicated or placebo)

SUMMARY:
The aim of the present randomized, double-blind study is to evaluate the effects of a vulvar, moisturizing, non-hormonal gel containing visnadine, ethil ximeninate, Coleus barbatus and Panicum miliaceum (TROFIS (R)), in women in the menacme, regarding the sexual response measured by the Female Sexual Function Index (FSFI) when compared to placebo.

DETAILED DESCRIPTION:
In this study, 60 sexually active (having a male partner, boyfriend or husband) female volunteers will be included. All patients will undergo gynecological evaluation of the vulvar area and the vaginal mucosa before and after the treatment, by means of visual inspection and speculum examination.

Volunteers will be requested to apply once a day, for four weeks, a small amount of gel to the dry area (vulva), followed by a gentle massage to promote the absorption of the product.

For the time of the study, volunteers will be asked not to change personal hygiene products, e.g., moisturizers, soaps, deodorants, etc. Volunteers will be instructed to fill out the "diary of use" with the dates of product application and notes about feelings of discomfort or subjective reactions, if any. In the final visit, volunteers will answer the FSFI questionnaire (see Annex 1). All variables in the questionnaire (comfort during sexual intercourse, hydration and softness of genital tissue) will undergo a descriptive analysis.

In the first moment of the study, patients will receive the FSFI (Female Sexual Function Index) questionnaire, self-applied and validated for the Portuguese language in Brazil (Thiel et al., 2008). Then, the estronization of external genital organs will be assessed by gynecological exam.

Patients will be randomly assigned to four groups: group A and B (A and B - 30 and 30 patients in the menacme, following the order defined by the computer-generated randomization list.

During the advertising process, patients will be interviewed by phone following the same chronological order of their contacts with the clinic and a medical evaluation will be scheduled.

The participants will be with age greater than 20 old, be in either the menacme (not pregnant). They will have complaints about sexual activity, an active sex life, and body mass index (BMI) equal to or less than 30. Through these criteria of inclusion and exclusion.

After collection of clinical history and gynecological anamnesis, these women will undergo a general physical examination and gynecological examination, oncotic cytology, and imaging examination of the endometrial thickness (transvaginal ultrasonography). With the exams results, the women will undergo another medical evaluation.

All participants will sign the Informed Consent Form (ICF). Patients in the menacme _ Group A and B (medicated or placebo) Biolab Farmaceutica (242 Rua das Olimpíadas, 3rd floor, Vila Olímpia/São Paulo - SP) will provide free of charge Trofis and placebo (inactive compound) gels. All tubes containing the gel will have the same shape and will be labeled with a batch number, which carries the information on the content, only known by Biolab. In this manner, blindness will be maintained for the entire study time, until the last patient finishes one month of treatment. Patients and the physician researcher will not know which gel contains the active component or to which group it belongs. The volunteers will apply once a day, for four weeks, a small amount of gel to the dry area (vulva), followed by a gentle massage to promote the absorption of the product.

In the end of the first month of treatment, patients will go to the clinic for a follow up to ensure treatment adherence and to evaluate potential adverse effects of the gel. After one month of treatment, patients will answer the FSFI questionnaire again, and will undergo a general clinical examination and gynecological examination of the external genital organs.

In the end of treatment and with results of complementary exams, patients will be instructed to continue attending the gynecological routine consultations in the Ginecologia Endócrina, outpatient clinic of EPM/UNIFESP.

ELIGIBILITY:
Inclusion Criteria:

- women with age greater than 20, in the menacme, with complaints about sexual activity.

Exclusion Criteria:

* body mass index (BMI) greater than 30

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 60 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2016-12-10 (Actual); Study Completion 2016-12-10 (Actual)

PRIMARY OUTCOMES:
improvement of sexual desire | 30 days
  The aim of the present randomized, double-blind study is to evaluate the effects of a vulvar, moisturizing, non-hormonal gel containing visnadine, ethil ximeninate, Coleus barbatus and Panicum miliaceum (TROFIS (R)), in women in the menacme, regarding the sexual response measured by the Female Sexual Function Index (FSFI) when compared to placebo.

IPD SHARING:
Plan to Share IPD: No
do not aplay